CLINICAL TRIAL: NCT05100056
Title: Effectiveness and Safety of Consolidative Brentuximab Vedotin (BV) Treatment Administered to Hodgkin's Lymphoma (HL) Patients That Had Undergone Autologous Stem Cell Transplant (ASCT). Prospective, Multicenter, Observational Study
Brief Title: A Study of Brentuximab Vedotin in Adults With Hodgkin's Lymphoma
Acronym: BV-MAZOVIA
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Brentuximab-5018
Record Dates: First submitted 2021-10-28; First posted 2021-10-29 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Hodgkin Lymphoma
Keywords: Drug Therapy
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HL Participants: BV Salvage Pre-ASCT: Participants diagnosed with HL who undergone or undergoing pre-ASCT BV salvage and continue with post-ASCT treatment will be observed prospectively over 24-month period after treatment cessation.
  Interventions: Other: No Intervention
- HL Participants: BV Consolidation Treatment Post-ASCT: Participants diagnosed with HL who undergone or undergoing post-ASCT BV consolidation treatment will be observed prospectively over 24-month period after treatment cessation.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The main aim is to check how effective BV is for treating adults with HL.

Study medication will be prescribed according to the clinic's standard practice.

Participants will visit the study clinic 5 times, once every 12 weeks. When study treatment has completed, a follow-up visit will be scheduled every 3 months during the first year and every 4-6 months during the next year.

DETAILED DESCRIPTION:
This is a prospective, observational study in participants with HL who underwent or are candidates for ASCT and receiving or will receive the standard treatment of BV. This study will assess the safety profile and effectiveness of BV in pre and post-ASCT in the real-world clinical practice.

The study will enroll approximately 70 participants.

The data will be collected and recorded in electronic case report forms (e-CRFs) in scope of National Drug Program (NDP). All the participants will be assigned to two observational cohorts:

* HL Participants: BV Salvage Pre-ASCT
* HL Participants: BV Consolidation Treatment Post-ASCT

This multi-center trial will be conducted in Poland. All participants will be followed up for 24 months. The overall duration of the study will be approximately 4.5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participant (aged greater than or equal to [>=18] years) that underwent or are candidates for ASCT and were enrolled in BV HL NDP receiving treatment according to the Summary of Product Characteristics for Adcetris and NDP.

Exclusion Criteria:

1. Currently participates or plans to participate in any interventional clinical trial.
2. Any other reason that, in the Investigator's opinion, makes the participant unsuitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with HL (previously enrolled in BV HL NDP) who underwent or are candidates for ASCT will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) as Assessed by Investigator | From initiation of BV treatment post-ASCT until disease progression or relapse, or death (up to 36 months)
  PFS will be assessed by investigator and defined as the time from the first dose of BV post ASCT until the first occurrence of disease progression or relapse, or death for any reason. Disease progression is at least a 50 percent (%) increase in the size of lesions, or the occurrence of new lesions. It will be analyzed using Kaplan-Meier method.

SECONDARY OUTCOMES:
Overall Survival (OS) | From initiation of BV treatment until death from any cause (up to 36 months)
  OS is defined as the time from initiation of therapy to death from any cause. It will be analyzed using Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (13):
- Poland (13):
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw, Dolnoslskie
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan, Greater Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy Oddzial w Krakowie, Krakow, Lesser Poland Voivodeship
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie, Krakow, Lesser Poland Voivodeship
  - Centrum Onkologii Ziemi Lubelskiej im. sw. Jana z Dukli, Lublin, Lublin Voivodeship
  - NU-MED Specjalistyczny Szpital Onkologiczny Tomaszow Mazowiecki, Tomaszow Mazowiecki, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne WUM, Warsaw, Masovian Voivodeship
  - Instytut Hematologii i Transfuzjologii, Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Gdansk, Pomeranian Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny im. Andrzeja Mieleckiego Slskiego Uniwersytetu Medycznego w Katowicach, Katowice, Slskie
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej MSWiA z Warminsko - Mazurskim Centrum Onkologii w Olsztynie, Olsztyn, Warmian-Masurian Voivodeship
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii, im. M. Kopernika w Lodzi, Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/618310f4eb0e19002afd69ff